CLINICAL TRIAL: NCT00113477
Title: A Single-Centre, Randomised Double-Blind Placebo-Controlled Study to Measure the Effect of Q10 and Selen Supplement on Muscular Adverse Events in Statin Therapy
Brief Title: The Effect of Q10 and Selen Supplement on Muscular Adverse Events in Statin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Pharma Nord (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 12004 - versjon 2; 2004-000797-31 (EudraCT); S-04159 (REK Sør); 11250 (NSD); 200500691 (SLV)
Record Dates: First submitted 2005-06-08; First posted 2005-06-09 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2008-09

CONDITIONS: Statin Therapy
Keywords: Q10; CoQ10; Coenzyme Q10; selen; selenoprotein; selenoproteins; adverse events; adverse effects; AE; myalgia; muscle; statin therapy; Indication for statin therapy
MeSH Terms: conditions — Myalgia | interventions — Tuberculin; Selenium

INTERVENTIONS:
Drug: Q10
Drug: Selen

SUMMARY:
The purpose of this study is to determine whether supplements of Q10 and Selen are effective in reducing muscular adverse events (AE) in statin therapy.

DETAILED DESCRIPTION:
Statins inhibit the synthesis of cholesterol by inhibiting the enzyme HMG-CoA reductase. The reduction of intracellular cholesterol leads to an increase in the number of LDL-receptors, and subsequent increased uptake and metabolism of LDL in the liver. Several large clinical trials have shown that the use of statins decreases morbidity and mortality in patients with risk factors for atherosclerotic disease. Unfortunately, 5% of statin users experience adverse events (mainly gastrointestinal [GI] and muscular).

Statins inhibit not only cholesterol synthesis, but also synthesis of other substances in the mevalonate pathway. Among these other substances are Q10 and selenoproteins.

It is well known that serum Q10 levels decrease during statin therapy, and that Q10 supplement inhibits this decrease. One study has shown reduction of Q10 in blood-platelets during statin therapy. Q10 is an important element in the mitochondrial respiratory chain. Depletion of Q10 leads to a reduction of high energy phosphates, anaerobe metabolism and mitochondrial dysfunction. This is suggested to be the cause of muscular adverse events in statin therapy. There are several reports of individuals relieved from muscular adverse effects after Q10 supplement, but no randomized, placebo controlled studies have been conducted.

Symptoms of selenoprotein deficiency are very similar to adverse events seen in statin therapy, but no clinical trials have been conducted to evaluate the effect of selen supplement on adverse effects of statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 - 75 years old
* Indication for statin
* Previous history of muscular AE on statin therapy.

Exclusion Criteria:

* If female, be of non-childbearing potential, i.e., post-menopausal (defined as >12 months since last menstrual period) or surgically sterilised, or using adequate barrier contraception if of childbearing potential.
* Previously serious muscular AE
* Patients taking drugs interacting with statins, and where these drugs cannot be stopped.
* Allergy against selen
* Liver or kidney failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction of muscular adverse events

SECONDARY OUTCOMES:
Muscular strength measured by SAAT
Correlation between serum Q10 concentration and adverse events
Serum Q10 concentration in comparison to subjects not experiencing AE
The effect of 12 weeks on Lipitor 10 mg x 1 on muscular function and AE

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Retterstøl, MD, Principal Investigator — Lipidklinikken, Rikshospitalet-Radiumhospitalet HF
Locations (1):
- Lipidklinikken, Rikshospitalet, Oslo, Oslo County, Norway